CLINICAL TRIAL: NCT03812887
Title: A Prospective, Open, Comparative, Multi-Centre Photopatch Test Study of Patients Suspected of Photoallergy to Organic Sunscreens and Topical Non-steroidal Anti-inflammatory Drugs Used Within Europe
Brief Title: Photopatch Test Study (POST Study)
Acronym: POST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mater Misericordiae University Hospital (Other)
Collaborators: European Association of Dermatology and Venerology (Unknown)
Responsible Party: Principal Investigator, Dr Nicola Ralph, Principal Investigator, Mater Misericordiae University Hospital
Other Study IDs: MaterMUH
Record Dates: First submitted 2019-01-03; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Photoallergy
MeSH Terms: conditions — Dermatitis, Photoallergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Photopatchtesting — Photopatchtesting to the sunscreen series and extended series, irradiated at both 24 and 48 hours
  Other Names: Patchtesting

SUMMARY:
In the year 2000, a group of specialists with an interest in contact dermatitis and photobiology/photophysics set up a taskforce under the umbrella of the European Society for Contact Dermatitis and the European Society for Photodermatology. This came about as a result of an awareness, that photopatch testing was under-used, there were inconsistencies in methodology and scoring of results, and there was a lack of up-to-date choice of test photoallergens. A consensus on the methodology of photopatch testing arose from this, although some inconsistencies on the methodology could not be solved and variations on the technique were accepted. Since then a European multicentre photopatch test study (EMCPPTS) was conducted in 30 clinics from 2008-2011. The EMCPPTS test agents comprised 19 UV absorbers, and 5 topical non-steroidal anti-inflammatory drugs available in Europe. More than 1,000 patients took part in this study that showed that ketoprofen and related chemicals and classical UV-filters were the main photoallergens.

Since then the taskforce have met again (2012) and on the basis of the results of the ECMPPTS, on previous publications reporting cases of photoallergic contact dermatitis, and on the presence or absence of these agents in consumer products within the European market or other accessible markets, 20 substances were chosen to form the baseline European photopatch test series. Fifteen additional substances were chosen to be included in the extended photopatch test series which may be used as an additional screen alongside patients' own product. Twenty-six other agents that are no longer produced or are no longer used in the European markets have been considered to be no longer relevant for regular photopatch testing and were removed.

It was suggested from this taskforce that the study should be repeated in approximately five years, as it is expected that new photoallergens will continue to emerge despite pre-marketing screening measures. Therefore members of this taskforce subsequently met in 2015, to discuss the aim of performing a very similar study, commencing in 2016. However, the investigators aim to focus specifically on methodology as in all previous studies a variety of methods of photopatch testing have been utilised. The investigators therefore aim to improve standardisation of this test. This agreed methodology will therefore enable better comparative studies in the future and hopefully encourage greater numbers of would-be users of this form of patch testing, as due to a previous level of uncertainty, many general dermatologists have been discouraged from using this technique.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine the frequency of photoallergic and allergic reactions to the most recently recommended battery of allergens used in photopatch testing in Europe.
2. To compare, within the same individual, photopatch tests results when the tests are irradiated at 24hr or 48hr in order to determine whether one or other time point is superior with respect to pick-up of relevant positive photoallergic reactions.

Secondary objective:

To evaluate whether use of an additional 7 day, late reading yields new and relevant reactions that increase the diagnostic capacity of photopatch testing.

The Chief Investigator (CI) for the study is Dr Niki Ralph, Dublin. All centres will each have a lead clinical dermatologist with a special interest in contact dermatitis or photobiology/photophysics. Many of these lead dermatologists have also been part of the taskforce in the last 16 years of studies/meetings surrounding this topic. Each lead dermatologist will have a multidisciplinary team at their centres and be regularly involved in patch/photopatch testing. Dundee will be the main co-ordinating site for the UK. Patients who are attending for patch/photopatch testing at each of these centres will be offered inclusion in the study. The primary indication for this form of testing includes dermatitis predominantly affecting exposed sites with or without a history of a reaction to sunscreen, anti-inflammatory drug or related agents and patients who are being investigated for photosensitivity diseases.

Participants & Recruitment Each patient will be given a participant information sheet (PIS. Appendix 1) and have at least 24 hours to read through this. They will also be given the opportunity to speak with a member of the research team, as contact details will be provided on the patient information sheet or they may wish to have any questions answered in person, during their consultation at the outpatient clinic, before they are invited to sign a standardised informed consent form (Appendix 2) prior to recruitment into the study. No study activity will take place until the patient has given written informed consent.

Methodology The patients will attend the clinic +/- two hours the same time each day (Table 1). Three sets of patch tests will be applied on 8mm Finn chambers to the back, or another body site if necessary, to facilitate the number of patchtest chambers required. One set for standard patch testing according to the International Contact Dermatitis Research Group (ICDDRG) criteria, one set of the agreed baseline 23 photoallergen series for irradiation at 24 hours and one set of the agreed baseline 23photoallergen series for irradiation at 48 hours, according to this study protocol. There is also an extended series of photoallergens. Patients may also be tested to this series, or only individual allergens from this series as deemed appropriate by their clinician, based on their medical history.

Randomisation Randomisation will be undertaken using a computer-generated randomisation sequence, taking into account which sites are applied for 24h/48h and which sites are irradiated/not irradiated.

Readings of the patch tests will be interpreted as follows (Table 1):

Table 1:

Day 0 (D0) Day 1 (D1) Day2 (D2) Day 3 (D3) (if feasible) Day 4 (D4) Day 7 (D7-late reading) (if feasible) Application of 2 identical sets of patch tests (PTs) Application of 3rd (final set) of identical PTs Removal of all PT's from the back. Reading of all sets of PT's Irradiation of 2 sets of PTs (24 & 48 hour irradiation) Immediate reading post irradiation Reading of PPTs (24 hour) Reading of PPTs (48 hour) Late reading of PPTs

Minimal Erythema Dose (MED) testing:

Patients who attend the photobiology centres may have a UVA MED test performed and recorded on the photopathc test recording sheet. (Appendix 3) For centres who are mainly contact allergy centres, they will use a standard dose of 5J/cm² UVA for patients who are not phototested or who have normal phototesting and those with moderate photosensitivity will be tested to 2.5J/cm² and those with severe photosensitivity will be tested using 1J/cm² UVA and this will be at the discretion of the study clinician at each centre.

Meter Calibration:

All UVA meters from the 13 included centres will be calibrated to ensure standardisation (prior to study use) in Dundee, Scotland, by Dr Ewan Eadie, Head of Scientific Services for Photobiology and Optical Radiation.

Assessor blinding:

This will be incorporated by all 13 centres, so that the assessor does not know which site is irradiated and also which are the 24 or 48 hour sites.

Assessing clinicians will be unaware of the ordering of the set of patches (24hr vs 48hr) allocated on the back. This will be achieved by the following:

Assessors will not be aware of the randomization schedule Assessors will not see the patches applied to the skin, but will only see the back/other areas once patches have been removed. The aim of this is to improve assessment robustness

Blinding will be broken in the event of a serious adverse event, or at study clinician request, due to clinical need. A copy of the open randomisation code will be stored in a locked cupboard in the clinic. This can be accessed in the event of an emergency requirement to break the blind.

Sunscreen series/Non-steroidal anti-inflammatory drug (NSAID) series:

All patients who agree to take part in the study will be offered testing to the entire sunscreen and NSAID series. However, topical NSAIDs are much more widely used in Continental Europe and, some patients, particularly in the UK, may not be aware of ever having been exposed to a topical NSAID. Patients who do not wish to be tested to NSAID's as they feel these may not be relevant to their individual situation can continue to participate in the study, however will only be tested to the sunscreen series +/- NSAIDs.

Inclusion Criteria

1. Aged 18 years and over
2. Referred for photodiagnostic testing or for patch testing for investigation of any of the following indications:

   Exposed-site dermatitis in summer months Any exposed site dermatitis History of reaction to sunscreen/NSAID or related agents Suspected or confirmed photosensitivity
3. Able to understand and comply with the restrictions and requirements of the study
4. Able to provide written informed consent

Exclusion Criteria

1. Unable to understand and comply with the restrictions and requirements of the study
2. Not able to give written informed consent
3. Recent sunburn/tan on back within 4 weeks of the planned photopatch testing
4. Systemic immunosuppressants, including oral corticosteroids (>10mg/day)
5. Active skin disease on back precluding testing.
6. Potent topical corticosteroid use to back within 5 days of planned recruitment and testing
7. Pregnancy or breastfeeding

Study Assessments During the study duration the data will be recorded onto a standardised photopatch test form (Appendix 3) and at the end of the study all forms will be collected from each individual study centre, under the direction of the local principal investigator (PI). These data will then be collated once all participants have been recruited.

The collective data will then undergo statistical analysis by the statistician at the Lead CI centre in Dublin.

Funding No external funding has been sought by the UK Investigators. The CI has secured minor funding from The City of Dublin Skin and Cancer Hospital Charity and from the EADV. Funding is available for reimbursement of participant travel expenses for up to the two extra visits (Up to 10 Euro per each visit) (Appendix 1)

Statistical Analysis The collective data will undergo statistical analysis by the statistician at the Lead CI centre in Dublin in order to investigate whether there is a difference between 24h versus 48h allergen application or whether addition of a late seven day reading increases the yield of relevant positive reactions. The investigators estimated, using Stata 14.1 (Stata Corp., Texas, 2016) that 189 completing subjects would give 90% power to detect as significant, at an alpha level of 0.05, a difference (assuming two-tailed testing) of 10% between within-subjects proportions of identified reactions at the 2 different randomly allocated durations of application of patches. This estimate was also based on the conservative assumption of an intraclass correlation coefficient of 0.01, in the absence of previous study data on which to base this estimate.

Feasibility This study's success is dependent on being able to acquire sufficient numbers of patients to undergo photopatch testing. Based on previous studies in this area, (from this taskforce) the investigators envisage that this will be possible but will require a lead coordinator (Dr Niki Ralph for Europe, Dr Sally Ibboston for UK) to oversee and conduct the study and be contactable on a regular basis by all centres to ensure the protocol is understood by the lead dermatologist and their team whom are involved in the study (doctors/nurses/physicists etc.) and to ensure that the exact protocol is being adhered to and the data are being collected and recorded according to the protocol.

The study centres who have agreed to be part of this study all have lead dermatologists who have a special interest in the areas of contact dermatitis, photobiology and photophysics and have participated in such studies in the past; hence we do not anticipate difficulties with acquiring large numbers of patients to undergo such testing.

Failure of the project could occur if patients did not attend on a regular basis for the interpretation of their test results. This is not envisaged by the group, as patients who attend for this form of patch testing are usually very enthusiastic about identifying the possible cause of their cutaneous reaction, hence compliance is usually very high. The addition of the late reading after a weekend break from the hospital may prove difficult for some patients, due to geographical location but is not a mandatory time-point for readings.

Data processing The data will be recorded on the standardised patchtest recording sheet for each individual patient participating in the study. The results will be stored in the patients' medical record in each individual centre and an anonymous copy will be sent to the P.I. Dr Niki Ralph. The photopatch recording sheets are anonymous. There will also be a master/consent log at each site linking the participant name to the number. Dr Ralph will record all data from the 13 centres on an Excel spreadsheet, which will be stored on a password encrypted, powered off computer, in a locked office. All data will be kept for the duration necessary to create publications and presentations at both national and international level, for approximately 5 years post completion of study.

The chief investigator reserves the right to conduct an audit of the informed consent process at each study site Insurance The coordinator for each centre is covered by their individual hospital indemnity and their own personal indemnity through an insurance provider.

Scientific Justification This study will contribute to the promotion of excellence in clinical care by investigation optimisation of an important diagnostic test in dermatology. It joins two special interest societies, the ESCD & ESPD who are collaborating to undertake a multi-centre study to define the prevalence of the most commonly encountered photoallergens in Europe and the most appropriate methodology for photopatch testing across Europe. The investigators aim to clarify the best method for photopatch testing to create a standard method, which could be a baseline study for all other European studies.

The investigators hope to act as advocates for patients and both consultant and trainee dermatologists and nurses and technologists; by involving them in a study, which will benefit the patients in the diagnosis of their skin condition and will assist in teaching and training of those involved in delivering photopatch test services. Publishing the findings in peer-reviewed journals and presenting at national and international dermatology meetings will be of major importance in dissemination of new knowledge obtained in the course this study and will contribute to the specialty of Dermatology by educating its members including those in sub-specialty groups.

Moreover, the correct identification of the causes of photoallergic dermatitis, namely in multi-centre studies, may give important indications to the institutions that deal with the safety of consumers and to the cosmetic/pharmaceutical industry in order to eliminate or reduce exposure to frequent photoallergens and, therefore, improve the quality of health of European citizens.

Conclusion Thus, at the conclusion of this study the investigators will have validated the European standard battery of photoallergens and be able to advise on the likely frequency of reactions to specific photoallergens and which are the most common culprits and defined the optimal methodology to use for photopatch testing, with either a 24h or 48h allergen irradiation time-point (or indeed if no difference is found then investigators will also be advised that either regime is appropriate). As a secondary objective if sufficient late 7 day reading data points are obtained, the investigators may be able to semi-quantitatively ascertain whether there is value in inclusion of this late time-point for reading photopatch tests.

Dissemination of Knowledge Gained The information gained from this study will be presented widely at National and International photobiology and dermatology meetings and will be published in peer-reviewed scientific journals.

References Bruynzeel et al., J Euro Acad Derm Venereol 2004; 18: 679-82 Kerr et al., Br J Dermatol 2012; 166: 1002-9 Goncalo et al., Contact Derm 2013; 68: 239-43 Bryden AM, Moseley H, Ibbotson et al. Photopatch testing of 1155 patients: results of the U.K. multicenter photopatch study group. Br J Dermatol, 2006; 155:737-747

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and over
2. Referred for photodiagnostic testing or for patch testing for investigation of any of the following indications:

   Exposed-site dermatitis in summer months Any exposed site dermatitis History of reaction to sunscreen/NSAID or related agents Suspected or confirmed photosensitivity
3. Able to understand and comply with the restrictions and requirements of the study
4. Able to provide written informed consent

Exclusion Criteria:

1. Unable to understand and comply with the restrictions and requirements of the study
2. Not able to give written informed consent
3. Recent sunburn/tan on back within 4 weeks of the planned photopatch testing
4. Systemic immunosuppressants, including oral corticosteroids (>10mg/day)
5. Active skin disease on back precluding testing.
6. Potent topical corticosteroid use to back within 5 days of planned recruitment and testing
7. Pregnancy or breastfeeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients attending the dermatology clinics for photopatch testing will be offerred inclusion into the study
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Record the frequency of photoallergic and allergic reactions to the most recently recommended battery of allergens used in photopatch testing in Europe | Two years
  Photopatchtesting to the most up to date Sunscreen series and extended series

SECONDARY OUTCOMES:
Compare within the same individual, photopatch tests results when the tests are irradiated at 24hr or 48hr in order to ascertain whether one or other time point is superior with respect to pick-up of relevant positive photoallergic reactions. | Two years
  Testing patients to both irradiation of the sunscreen series at 24 and 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Only the final result (total figures/statistics) will be shared with other researchers, data is anonymised and other centres involved in the study will only have final data not each other centres individual results